CLINICAL TRIAL: NCT06556953
Title: Development and Validation of Machine Learning Models to Evaluate the Postoperative Venous Thromboembolism Risk of Cervical Cancer Patients in China
Brief Title: Evaluating the Risk of Postoperative Venous Thromboembolism in Cervical Cancer Patients
Status: Completed | Type: Observational
Sponsor: Haike Lei (Other)
Responsible Party: Sponsor-Investigator, Haike Lei, director, Chongqing University Cancer Hospital
Organization: Chongqing University Cancer Hospital (Other)
Other Study IDs: CZLS2023337-A
Record Dates: First submitted 2024-08-06; First posted 2024-08-16 (Actual); Last update posted 2024-08-16 (Actual); Status verified 2024-08

CONDITIONS: Venous Thromboembolism
Keywords: machine learning; postoperative VTE; cervical cancer
MeSH Terms: conditions — Venous Thromboembolism; Uterine Cervical Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The aim of this study is to develop a machine learning model to accurately predict the risk of venous thromboembolism in patients with cervical cancer after surgery.

DETAILED DESCRIPTION:
Venous thromboembolism (VTE) is a common and life-threatening complication in patients with cervical cancer following surgery. The objective of this study is to develop a machine learning model with the potential to predict the risk of VTE in these patients postoperatively. We plan to employ partial dependence (PD) curves, breakdown (BD) curves, Ceteris-paribus (CP), and SHapley additive exPlanations (SHAP) values for a comprehensive analysis. The goal is to explore how different machine learning algorithms can be utilized as tools for personalized postoperative VTE risk assessment in cervical cancer patients.

ELIGIBILITY:
Inclusion Criteria:

* Confirmation of cervical cancer through pathological examination.
* Receipt of surgical treatment for cervical cancer at Chongqing University Cancer Hospital in China.
* Provision of comprehensive case information.

Exclusion Criteria:

* Patients under the age of 18.
* History of VTE caused by other reasons before surgery.
* Secondary cervical cancer or accompanying primary malignant tumor.

Ages: 20 Years to 89 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Our data was collected from electronic case of the cervical cancer patients who underwent surgical treatment at the Cancer Hospital affiliated with Chongqing University between January 2019 and December 2022
Sampling Method: Non-Probability Sample
Enrollment: 1174 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Whether the patient has developed VTE is determined based on the diagnostic criteria in the "Guidelines for the Prevention and Treatment of Tumor-Associated Venous Thromboembolism (2019 Edition)." | December 31, 2023
  The diagnosis of VTE primarily includes the diagnosis of DVT and PE. According to the guidelines, DVT is diagnosed using venous compression ultrasound or venography, while PE is diagnosed using CT pulmonary angiography (CTPA) or nuclear lung ventilation/perfusion imaging.

CONTACTS AND LOCATIONS:
Locations (1):
- Chongqing University Cancer Hospital, Chongqing, Chongqing Municipality, China